CLINICAL TRIAL: NCT03298230
Title: A Pilot Randomised Controlled Trial of REmotely SuPervised Exercise Training for Patients With Peripheral Arterial Disease: The RESPECT-PAD Trial
Brief Title: The RESPECT-PAD Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Charles McCollum, Professor of Surgery, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 224506
Record Dates: First submitted 2017-09-21; First posted 2017-10-02 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REmotely SuPervised Exercise Training (Experimental): 12- week home based exercise programme consisting of bi-weekly, hourly sessions at the time and place of the participant's choosing. They will wear a fitness tracker which will automatically upload their exercise data to an online platform which can be monitored by the research team and used to provide additional motivation.
  Interventions: Behavioral: REmotely SuPervised Exercise Training
- Supervised Exercise Training (Active Comparator): As per NICE guidance. 12 week, bi-weekly, one hour sessions of supervised exercise training.
  Interventions: Behavioral: Supervised Exercise Training

INTERVENTIONS:
Behavioral: REmotely SuPervised Exercise Training — As described in the Arms section.
  Arms: REmotely SuPervised Exercise Training
Behavioral: Supervised Exercise Training — As described in the Arms section.
  Arms: Supervised Exercise Training

SUMMARY:
Peripheral arterial disease affects around 25% of the UK population aged over 55. Left untreated it can lead to debilitating pain, gangrene, amputation and death. It most commonly affects the lower limbs and in the earlier stages of the disease patients can present with a symptom known as intermittent claudication; pain felt in the legs which stops the patient from walking past a certain distance. Current National Institute for Healthcare and Excellence (NICE) guidelines recommend Supervised Exercise as first line treatment for patients with peripheral arterial disease presenting with intermittent claudication. Supervised exercise employs behaviour changing techniques which enable the patient to modify their lifestyles, improving their claudication symptoms, quality of life and reducing their cardiovascular risk. Despite this treatment being significantly more cost-effective than often employed complex endovascular management, most institutions don't offer such programmes citing lack of resources and compliance from clinicians and patients alike.

The investigators propose a more cost-effective, resource-savvy solution in the form of REmotely SuPervised ExerCise Training (RESPECT). This allows the patient to exercise in the convenience of their own home, at a time of their choosing but still be supervised via fitness tracker technology and an online fitness platform. This randomised controlled trial will attempt to prove its' effectiveness in increasing claudication distance, improving functional ability, decreasing cardiovascular risk and improving quality of life whilst being more cost-effective than the currently recognised national first line treatment. This trial has the potential to revolutionise the management of patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to undertake supervised or home-based exercise training aged between 40 and 85
2. Positive Edinburgh questionnaire for intermittent claudication (APPENDIX H)
3. Proven peripheral arterial disease on diagnostic imaging
4. Ankle Brachial Pressure Index (ABPI) <0.9
5. Fontaine Classification (APPENDIX I) of PAD Stage II
6. Conservative management plan agreed for by Consultant Vascular Surgeon.

Exclusion Criteria:

1. Critical limb ischaemia
2. Asymptomatic peripheral arterial disease
3. Ambulation limited by co-morbid condition other than claudication:

   Severe coronary artery disease, angina pectoris, chronic lung disease, neurological disorder, arthritis, amputation
4. Contraindication to exercise training (AHA guidelines):71 acute MI (within 1 week), unstable angina, uncontrolled cardiac arrhythmias causing symptoms or haemodynamic compromise, active endocarditis, symptomatic severe aortic stenosis, acute pulmonary embolus, acute noncardiac disorder than may be aggravated by exercise such as infection, thyrotoxicosis, acute myocarditis, known physical disability that would preclude safe and adequate testing, known thrombosis of the lower limb, known left main stem coronary stenosis, moderate stenotic valvular heart disease, pulmonary hypertension, hypertrophic cardiomyopathy, atrio-ventricular block.
5. Psychiatric disorder precluding them from consenting for research and/or exercise training
6. Arterial reconstruction in the previous 12 months or planned within the next 6 months.
7. Recent or upcoming major surgery (within 3 months)
8. Unwilling or unable to attend/perform exercise training
9. Non-atherosclerotic cause of PAD
10. Other significant medical problems which impact on the patient's ability to complete a 12-week exercise programme, which could include:

malignancy, chronic renal disease, chronic liver disease or anaemia, active substance abuse, dementia

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Absolute Claudication Distance | At 12 weeks
  Measured using a G-protocol on treadmill testing

SECONDARY OUTCOMES:
Absolute Claudication Distance | 6 months and 1 year.
  Measured using a G-protocol on treadmill testing
Initial Claudication Distance | 12 weeks, 6 months and one year
  Measured using a G-protocol on treadmill testing
Health-related Quality of Line | 12 weeks, 6 months and one year
  Measured using the Medical Outcomes SF36v2 Questionnaire
Cardiovascular Risk Factors | 12 weeks, 6 months and one year
  Measured by calculating change in waist circumference and BMI
Cost | 12 weeks, 6 months and one year
  Measured by the cost of the interventions in each group, including resource and staffing costs. Also includes any unplanned admissions and procedures carried out due to a complication of the disease of interest
Habitual physical activity levels | 12 weeks, 6 months and one year
  As measured by the physical activity scale for the elderly questionnaire.
Adherence | 12 weeks, 6 months and one year
  As measured by using the amount of exercise in minutes performed over the 12 weeks, divided by the number of minutes of exercise prescribed x100

IPD SHARING:
Plan to Share IPD: Undecided